CLINICAL TRIAL: NCT02065154
Title: Phase II Clinical Trial of the Use of Post-Transplant Cyclophosphamide for Graft Versus Host Disease (GvHD) Prophylaxis Following Matched Unrelated Donor (MUD) and Mismatched Unrelated Donor (MMUD)Hematopoietic Stem Cell Transplant (HSCT)
Brief Title: Post Transplant Cyclophosphamide (Cytoxan) for GvHD Prophylaxis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Omer Jamy, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UAB 1286
Record Dates: First submitted 2013-11-05; First posted 2014-02-17 (Estimated); Results first posted 2022-06-15 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Leukemia; Lymphoma; Myelodysplastic Syndrome; Myelofibrosis; Severe Aplastic Anemia; Allogeneic Transplant
Keywords: acute myeloid leukemia; AML; acute lymphoblastic leukemia; ALL; chronic myeloid leukemia; CML; chronic lymphocytic leukemia; CLL; non-Hodgkin lymphoma; NHL; Hodgkin lymphoma; HL; myelodysplastic syndrome; MDS; myelofibrosis; severe aplastic anemia
MeSH Terms: conditions — Leukemia; Lymphoma; Myelodysplastic Syndromes; Primary Myelofibrosis; Anemia, Aplastic; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin; Hodgkin Disease | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cyclophosphamide (Cytoxan) (Experimental): Cyclophosphamide (Cytoxan)
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Cyclophosphamide
  Other Names: Cytoxan

SUMMARY:
The main purpose of this study is to assess the effects of cyclophosphamide (cytoxan) in the post transplant setting to prevent onset of acute graft-versus-host disease (GVHD). The primary objective is to determine the incidence of grade II-IV acute GVHD following Allogeneic (allo) Hematopoeitic Cell Transplant (HCT) using post-transplant cyclophosphamide (cytoxan) for patients with human leukocyte antigen (HLA) matched unrelated (MUD) and mismatched unrelated (MMUD) donors. Other objectives for this study will be the determination of disease-free survival (DFS) and overall survival (OS) following allo HCT and assess the safety of post-transplant cyclophosphamide (cytoxan) for MUD and MMUD transplantation. Disease recurrence and time to recurrence in patients receiving post-transplant cyclophosphamide compared to historical control without post-transplant cyclophosphamide (cytoxan) will also be evaluated. Other objectives will be to determine the time of onset, severity, responsiveness to treatment, organs involved of acute and chronic GVHD as well as observation of Immune Reconstitution over time.

DETAILED DESCRIPTION:
he main purpose of this study is to assess the effects of cyclophosphamide (cytoxan) in the post transplant setting to prevent onset of acute graft-versus-host disease (GVHD). The primary objective is to determine the incidence of grade II-IV acute GVHD following Allogeneic (allo) Hematopoeitic Cell Transplant (HCT) using post-transplant cyclophosphamide (cytoxan) for patients with human leukocyte antigen (HLA) matched unrelated (MUD) and mismatched unrelated (MMUD) donors. Other objectives for this study will be the determination of disease-free survival (DFS) and overall survival (OS) following allo HCT and assess the safety of post-transplant cyclophosphamide (cytoxan) for MUD and MMUD transplantation. Disease recurrence and time to recurrence in patients receiving post-transplant cyclophosphamide compared to historical control without post-transplant cyclophosphamide (cytoxan) will also be evaluated. Other objectives will be to determine the time of onset, severity, responsiveness to treatment, organs involved of acute and chronic GVHD as well as observation of Immune Reconstitution over time.

ELIGIBILITY:
Inclusion Criteria:

* Disease Criteria: patients must meet diagnostic criteria of acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), chronic myeloid leukemia (CML), chronic lymphocytic leukemia (CLL), non-Hodgkin lymphoma (NHL), Hodgkin lymphoma (HL), myelodysplastic syndrome (MDS), myelofibrosis, or severe aplastic anemia. Patients will be allowed on study if they are deemed eligible for allo HCT regardless of remission status.
* Age Criteria: 19 to 65 years in age.
* Organ Function Criteria: All organ function testing should be done within 28 days of study registration.
* Cardiac: Left ventricular ejection fraction (LVEF) ≥ 50% by MUGA (Multi Gated Acquisition) scan or echocardiogram.
* Pulmonary: FEV1 (Forced expiratory volume in 1 second) and FVC (Forced vital capacity) ≥ 50% predicted, DLCO (diffusing capacity of the lung for carbon monoxide) (corrected for hemoglobin) ≥ 50% of predicted.
* Renal: The estimated creatinine clearance (CrCl) must be equal or greater than 60 mL/min/1.73 m2 as calculated by the Cockcroft-Gault Formula:

CrCl=(140-age) x weight(kg) x 0.85 (if female)/72 x serum creatinine (mg/dL)

* Hepatic:

  * Serum bilirubin 1.5 upper limit of normal (ULN)
  * Aspartate transaminase (AST)/alanine transaminase (ALT) 2.5 ULN
  * Alkaline phosphatase 2.5 ULN
* Performance status: Karnofsky ≥ 70%.,
* Patient must be informed of the investigational nature of this study in accordance with institutional and federal guidelines and have the ability to provide written informed consent prior to initiation of any study-related procedures, and ability, in the opinion of the principal investigator, to comply with all the requirements of the study.
* Patient has a suitable and willing HLA-8/8 matched or 6/8 mismatched (at one allele) unrelated donor identified.

Exclusion Criteria:

* Non-compliant to medications.
* No appropriate caregivers identified.
* HIV1 (Human Immunodeficiency Virus-1) or HIV2 positive
* Uncontrolled medical or psychiatric disorders.
* Uncontrolled infections, defined as positive blood cultures within 72 hours of study entry, or evidence of progressive infection by imaging studies such as chest CT scan within 14 days of registration.
* Active central nervous system (CNS) leukemia.
* Preceding allogeneic HSCT.
* Pregnancy or Breastfeeding.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-08-27 (Actual); Primary Completion 2022-04 (Actual); Study Completion 2022-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Racquel D Innis-Shelton, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Bone Marrow Transplantation and Cellular Therapy Program, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Jamy O, Innis-Shelton R, Bal S, Paluri R, Salzman D, Di Stasi A, Costa L, Meredith R, Lamb L, Minagawa K, Mineishi S, Saad A. Phase II clinical trial of one dose of post-transplant cyclophosphamide for graft versus host disease prevention following myeloablative, peripheral blood stem cell, matched-unrelated donor transplantation. Am J Hematol. 2021 Oct 1;96(10):E396-E398. doi: 10.1002/ajh.26296. Epub 2021 Jul 31. No abstract available. PMID 34288026
- See also: UAB Bone Marrow Transplantation and Cell Therapy Program — http://www.uab.edu/medicine/bonemarrow/

RESULTS

PARTICIPANT FLOW:
Groups:
- Cyclophosphamide (Cytoxan): Cyclophosphamide (Cytoxan)
  Cyclophosphamide
Period: Overall Study
Arm/Group | Cyclophosphamide (Cytoxan)
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment: Cyclophosphamide (Cytoxan)
  Cyclophosphamide
Arm/Group | Treatment
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Grade II-IV Acute GVHD
Description: To calculate the percentage of patients developing graft versus host disease, grade II-IV, in the first 100 days after transplant
Time Frame: Till 100 days post transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 39
percentage of participants | 30 [15.2 to 40.1]

2. Secondary Outcome: Overall Survival
Description: What percentage of participants were alive at a certain time point after transplant
Time Frame: 2 Year Post Transplant
Measure: Number; unit: percentage of participants
Arm/Group | Cyclophosphamide (Cytoxan)
Number analyzed (Participants) | 39
percentage of participants | 51

3. Secondary Outcome: Disease-free Survival
Description: What percentage of participants did not have relapse of disease after transplant
Time Frame: 1 Year Post-transplant
Measure: Number; unit: percentage of participants
Arm/Group | Cyclophosphamide (Cytoxan)
Number analyzed (Participants) | 39
percentage of participants | 46.15

4. Secondary Outcome: Regimen Related Toxicity
Description: Number of toxicities experienced by the patients in the study
Time Frame: 100 Days Post Transplant
Measure: Number; unit: Number of toxicities
Arm/Group | Cyclophosphamide (Cytoxan)
Number analyzed (Participants) | 39
Number of toxicities | 6

5. Secondary Outcome: Relapse Rate
Description: What percentage of participants relapsed
Time Frame: 2 years post-transplant
Measure: Number; unit: percentage of participants
Arm/Group | Cyclophosphamide (Cytoxan)
Number analyzed (Participants) | 39
percentage of participants | 21

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Cytoxan: Patients getting cytoxan
Arm/Group | Cytoxan
All-Cause Mortality (participants affected / at risk) | 19/39
Serious Adverse Events (participants affected / at risk) | 8/39
Other Adverse Events (participants affected / at risk) | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cytoxan (N=39)
Tamponade (Cardiac disorders) | 1 (1)
AKI (Renal and urinary disorders) | 2 (2)
Resp distress (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 1 (1)
Serious infection (Hepatobiliary disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-22): https://cdn.clinicaltrials.gov/large-docs/54/NCT02065154/Prot_SAP_000.pdf
  • Informed Consent Form (2015-03-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT02065154/ICF_001.pdf